CLINICAL TRIAL: NCT00652899
Title: MT2007-19R: WCC #53 Allogeneic Natural Killer Cells in Patients With Recurrent Ovarian Cancer, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Allogeneic Natural Killer Cells in Patients With Recurrent Ovarian Cancer, Fallopian Tube, and Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to toxicity
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS138; UMN-MT2007-19R (Other: Blood and Marrow Transplantation Program); UMN-WCC-53 (Other: Women's Cancer Center, U of M); UMN-0712M23462 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Allopurinol; Cyclophosphamide; fludarabine phosphate; fludarabine; Whole-Body Irradiation; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Body Irradiation (Experimental): This group includes patients that received all chemotherapy, infusion of natural killer (NK) cells and total body irradiation per protocol.
  1. Allopurinol 300 mg by mouth daily (unless known allergy) before beginning chemotherapy and continuing through day 14 post NK cell infusion. 2. Cyclophosphamide 60 mg/m^2 on Days 4 and 5 preceding NK cell infusion. 3. Fludarabine phosphate 25 mg/m^2 on Days 6 through 2 preceding NK cell infusion. 4. Radiation: total-body irradiation 200 cGy Day 1 preceding NK cell infusion. 5. Allogeneic natural killer cells- Given day 0 - dose of 1.5-8.0 * 10^7/kg. 6. Aldesleukin 10 million units 3 times/week for a total of 6 doses beginning Day 0.
  Interventions: Biological: Allopurinol; Drug: Cyclophosphamide; Drug: Fludarabine phosphate; Radiation: total-body irradiation; Biological: Allogeneic natural killer cells; Biological: Aldesleukin
- No Total Body Irradiation (Experimental): This group includes patients that received chemotherapy and infusion of natural killer cells, but did not receive total body irradiation.
  1. Allopurinol 300 mg by mouth daily (unless known allergy) before beginning chemotherapy and continuing through day 14 post NK cell infusion. 2. Cyclophosphamide 60 mg/m^2 on Days 4 and 5 preceding NK cell infusion. 3. Fludarabine phosphate 25 mg/m^2 on Days 6 through 2 preceding NK cell infusion. 4. Allogeneic natural killer cells- Given day 0 - dose of 1.5-8.0 * 10^7/kg. 5. Aldesleukin 10 million units 3 times/week for a total of 6 doses beginning Day 0.
  Interventions: Biological: Allopurinol; Drug: Cyclophosphamide; Drug: Fludarabine phosphate; Biological: Allogeneic natural killer cells; Biological: Aldesleukin

INTERVENTIONS:
Biological: Allopurinol — All patients are to receive allopurinol 300 mg PO daily (unless known allergy) before beginning chemotherapy and continuing through day 14 post natural killer cell infusion.
  Other Names: Zyloprim
Drug: Cyclophosphamide — 60 mg/m^2 on Days 4 and 5 preceding natural killer cell infusion.
  Other Names: Cytoxan
Drug: Fludarabine phosphate — 25 mg/m^2 on Days 6 through 2 preceding natural killer cell infusion.
  Other Names: Fludarabine
Radiation: total-body irradiation — 200 cGy Day 1 preceding natural killer cell infusion.
  Other Names: TBI
  Arms: Total Body Irradiation
Biological: Allogeneic natural killer cells — Given day 0 - dose of 1.5-8.0 * 10^7/kg
  Other Names: related donor haploidentical allogenic cell infusion
Biological: Aldesleukin — 10 MU 3 times/week for a total of 6 doses beginning Day 0
  Other Names: IL-2; Interleukin-2

SUMMARY:
RATIONALE: Giving chemotherapy, such as cyclophosphamide and fludarabine, and total-body irradiation before a donor natural killer cell infusion helps stop the growth of tumor cells. It also helps stop the patient's immune system from rejecting the donor's natural killer cells. Aldesleukin may stimulate the natural killer cells to kill ovarian, fallopian tube, or primary peritoneal cancer cells. Treating the donor natural killer cells with aldesleukin may help the natural killer cells kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving laboratory-treated donor natural killer cells together with aldesleukin works when given after cyclophosphamide, fludarabine, and total-body irradiation in treating patients with recurrent and/or metastatic ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the in vivo expansion of an infused allogeneic natural killer (NK) cell product following a preparative regimen comprising cyclophosphamide, fludarabine phosphate, and total-body irradiation in treating patients with recurrent and/or metastatic ovarian, fallopian tube, or primary peritoneal cancer.

Secondary

* To characterize the quantitative and qualitative toxicities of this treatment regimen.
* To estimate disease response (complete or partial response) or clinical benefit (stable disease for > 6 months) as measured by Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
* To estimate time to progression and overall survival.
* To estimate the association between clinical response and donor/recipient KIR ligand matching status.

Tertiary

* To evaluate immune activation of the in vivo expanded haploidentical allogeneic NK cells and its effect on the immune system.

OUTLINE:

* Preparative regimen: Patients receive fludarabine phosphate IV on days 6 to 2 preceding natural killer (NK) cell infusion and cyclophosphamide IV on days 5 and 4 preceding NK cell infusion. Patients also undergo total-body irradiation on day 1 preceding NK cell infusion.
* Allogeneic natural killer (NK) cell administration and aldesleukin: Patients receive aldesleukin-activated haploidentical allogeneic NK cells intravenously (IV) on day 0. Beginning 4-6 hours after allogeneic NK cell infusion, patients receive aldesleukin subcutaneously (SC) 3 times a week for 6 doses.

Patients achieving any initial response (complete or partial response) or a clinical benefit (stable disease for > 6 months) who progress after 6 months may receive 1 re-treatment course as above.

Blood samples are collected at baseline, on days 0, 7, 14, and 28, and then at 2 and 3 months post NK cell infusion for cytokine measurements, immunophenotyping, functional analyses, and testing for persistence of donor cells.

After completion of study treatment, patients are followed periodically for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent ovarian cancer, fallopian tube, or primary peritoneal cancer who meets the following criteria:
* Measurable disease (≥ 1 cm) per Response Evaluation Criteria for Solid Tumors (RECIST) - patients with bone as their only site of metastatic disease will not be eligible
* Progression on or failure to respond to at least 2 salvage chemotherapy regimens (2 regimens given for disease recurrence) for recurrent/metastatic ovarian, fallopian tube, or primary peritoneal cancer
* If history of brain metastases, stable for at least 3 months after treatment - A brain computed tomography (CT) scan will only be required in subjects with known brain metastases at the time of enrollment or in subjects with new clinical signs or symptoms suggestive of brain metastases.
* Available related HLA-haploidentical natural killer (NK) cell donor (by at least class I serologic typing). If biologic parents or siblings are available, can proceed with work-up of subject prior to return of human leukocyte antigen (HLA) typing results.
* Age 18 years or older
* Gynecology Oncology Group (GOG) performance status 0 or 1
* Adequate organ function as determined by the following criteria within 14 days of study enrollment:

  * Bone marrow: platelets ≥ 80,000 x 10^9/L and hemoglobin ≥ 9g/dL, unsupported by transfusions; absolute neutrophil count (ANC) ≥ 1000 x 10^9/L, unsupported by granulocyte-colony stimulating factor (G-CSF) or granulocyte macrophage-colony stimulating factor (GM-CSF)
  * Renal function: creatinine (Cr) ≤ 2.0 mg/dL
  * Liver function: aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase < 5 times upper limit of institutional normal
  * Cardiac: Left ventricular ejection fraction >40%
  * Pulmonary function: > 50% corrected Carbon Monoxide Diffusing Capacity (DLCO) and Forced expiratory volume in one second (FEV1), if presence of pleural effusion due to metastatic disease >40% corrected DLCO and FEV1 acceptable.
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to Day 0
* Voluntary written informed consent signed before performance of any study related procedure not part of normal medical care.

Exclusion Criteria:

* Pregnant or lactating - The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active infection - subjects must be afebrile, off antibiotics, and with no uninvestigated radiologic lesions (infiltrates or lesions with negative cultures or biopsies are allowed).

Human anti-mouse antibody (HAMA) monitoring: All subjects will be questioned about prior exposure to antibody therapy (including OKT3, Rituximab, Trastuzumab, etc). Responses will be recorded and reported to the FDA as part of the annual report. For subjects with no prior antibody therapy exposure, no further action will be taken. For subjects who have received previous antibody therapies 10 ml of serum (red top tube) will be drawn before starting therapy and banked per section 8.1. The presence of HAMA will not exclude a patient from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Geller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients did not receive all of study treatment per protocol.
Groups:
- All Patients Enrolled: This group includes all patients consented to participate in this study.
Period: Overall Study
Arm/Group | All Patients Enrolled
Started | 14
Completed | 12
Not Completed | 2
Not completed — Death | 1
Not completed — Treating physician decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients Enrolled
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With In Vivo Expansion of Infused Allogeneic Natural Killer (NK) Cell Product
Description: Detection of an absolute donor derived cell count of > or = 100 cells/mL after NK cell infusion.
Time Frame: Day 12-14
Measure: Number; unit: Patients
Groups:
- Ovarian/Fallopian Tube/Peritoneal Cancer Patients: This group includes patients with recurrent ovarian, fallopian tube or primary peritoneal cancer who received at least one dose of chemotherapy (cyclophosphamide 60 mg/m^2 and fludarabine 25 mg/m^2 for 2 doses, and aldesleukin 10 million units for 6 doses), infusion of natural killer cells (1.5-8.0 * 10^7 kg) and/or total body irradiation per protocol (200 Gy on Day 1 preceding natural killer cell infusion).
Arm/Group | Ovarian/Fallopian Tube/Peritoneal Cancer Patients
Number analyzed (Participants) | 12
Patients | 0

2. Secondary Outcome: Number of Patients Per Disease Response
Description: Response Evaluation Criteria in Solid Tumors (RECIST) criteria: Complete Response (CR)-Disappearance of all target lesions (TL); Partial Response (PR)-< or = 30% decrease in the sum of the longest diameter (LD) of TL, reference baseline sum LD; Stable Disease (SD)-Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference the smallest sum LD since the treatment started; Progressive Disease (PD)- < or = 20% increase in the sum of the LD of TL, reference the smallest sum LD recorded since treatment started or appearance of < or = 1 new lesion.
Time Frame: 1 Month After Natural Killer Cell Infusion (Day 30)
Population: Includes 12 patients that completed treatment per protocol criteria.
Measure: Number; unit: Patients
Groups:
- No Total Body Irradiation: This group includes patients with recurrent ovarian, fallopian tube or primary peritoneal cancer who received at least one dose of chemotherapy (cyclophosphamide 60 mg/m^2 and fludarabine 25 mg/m^2 for 2 doses, and aldesleukin 10 million units for 6 doses), infusion of natural killer cells (1.5-8.0 * 10^7 kg) and no total body irradiation.
- Total Body Irradiation: This group includes patients with recurrent ovarian, fallopian tube or primary peritoneal cancer who received at least one dose of chemotherapy (cyclophosphamide 60 mg/m^2 and fludarabine 25 mg/m^2 for 2 doses, and aldesleukin 10 million units for 6 doses), infusion of natural killer cells (1.5-8.0 * 10^7 kg) and total body irradiation (200 Gy on Day 1 preceding natural killer cell infusion).
Arm/Group | No Total Body Irradiation | Total Body Irradiation
Number analyzed (Participants) | 7 | 5
Patients
  Complete Response | 0 | 0
  Partial Response | 2 | 1
  Stable Disease | 4 | 4
  Progressive Disease | 1 | 0

3. Secondary Outcome: Median Number of Days to Progression
Description: Median number of days from first date of treatment to date of disease progression (appearance of new metastatic lesions or objective tumor progression). Defined by computated tomography (CT) imaging based on Response Evaluation Criteria In Solid Tumors (RECIST): Progressive Disease (PD) > or = 20% increase in sum of all target or any new lesions.
Time Frame: From date of first treatment to disease progression
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | No Total Body Irradiation | Total Body Irradiation
Number analyzed (Participants) | 7 | 5
Days | 107 [8 to 200] | 90 [69 to 130]

4. Secondary Outcome: Median Overall Survival Number of Days Patients Alive After Treatment
Description: Median number of days patients alive from date of treatment to date of death or date of last follow-up if censored.
Time Frame: From first date on-study (treatment) to date of death
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Total Body Irradiation: This group includes patients that received chemotherapy, infusion of natural killer cells and total body irradiation per protocol.
- No Total Body Irradiation: This group includes patients that received chemotherapy, infusion of natural killer cells and no total body irradiation per protocol.
Arm/Group | Total Body Irradiation | No Total Body Irradiation
Number analyzed (Participants) | 5 | 7
Days | 171.5 [144 to 199] | 291 [8 to 301]

ADVERSE EVENTS:
Time Frame: Serious adverse events were monitored through the follow-up period; death was followed for up to 2 years after Day 1 treatment.
Description: Adverse event collection for the purposes of this study focused on targeted adverse events and unexpected adverse events at specific time points in relation to the NK cell infusion and post infusion IL-2 injections.
Arm/Group | All Patients Enrolled
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Enrolled (N=14)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constitutional symptoms (General disorders) | 1 (2)
Death - disease progression NOS (General disorders) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) — immune hemolytic anemia, drug-related hemolysis
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infection - febrile neutropenia (Infections and infestations) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Pain - abdomen NOS (Gastrointestinal disorders) | 1 (1)
Tumor lysis syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Enrolled (N=14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (23)
Fever (General disorders) | 12 (42)
Chills (General disorders) | 12 (44)
Hypertension (Cardiac disorders) | 1 (8)
Fatigue (General disorders) | 13 (115)
Edema (Blood and lymphatic system disorders) | 6 (29)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (17)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 11 (58)
Rash (Skin and subcutaneous tissue disorders) | 11 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (18)
Vomiting (Gastrointestinal disorders) | 11 (30)
Nausea (Gastrointestinal disorders) | 12 (80)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (28)
Sweats (Skin and subcutaneous tissue disorders) | 10 (27)
Positive blood culture with fever (Blood and lymphatic system disorders) | 2 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Endpoint for association of clinical benefit response with donor/recipient KIR ligand matching status is not evaluable due to 0 complete responders.

Correlative laboratory objectives are irrelevant due to ineffectiveness of study regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No